CLINICAL TRIAL: NCT07242846
Title: EFFECT OF INTRAARTICULAR TRIAMCINOLONE HEXACETONIDE AND BETAMETHASONE ON INTRAOCULAR PRESSURE: A PROSPECTIVE RANDOMIZED STUDY
Brief Title: EFFECT OF INTRAARTICULAR TRIAMCINOLONE HEXACETONIDE AND BETAMETHASONE ON INTRAOCULAR PRESSURE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Hilal YAĞAR, Assist. Prof, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025/55
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Knee Osteoarthritis (Knee OA); Intraocular Pressure
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — betamethasone dipropionate, betamethasone sodium phosphate drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Betamethasone (Active Comparator): Intraarticular betamethasone group
  Interventions: Drug: Diprospan
- Triamcinolone Hexacetonide (Active Comparator): Intraarticular triamcinolone hexacetonide
  Interventions: Drug: artropan

INTERVENTIONS:
Drug: Diprospan — Single intra-articular injection of betamethasone into the affected knee joint at baseline as part of routine care for symptomatic early-stage knee osteoarthritis. No additional intra-articular corticosteroid injections are given during the follow-up period.
  Arms: Betamethasone
Drug: artropan — Single intra-articular injection of triamcinolone hexacetonide into the affected knee joint at baseline as part of routine care for symptomatic early-stage knee osteoarthritis. No additional intra-articular corticosteroid injections are given during the follow-up period
  Arms: Triamcinolone Hexacetonide

SUMMARY:
This study is being done to find out whether two commonly used corticosteroid injections for knee osteoarthritis - betamethasone and triamcinolone hexacetonide - have different effects on eye pressure (intraocular pressure). Adults with painful early-stage knee osteoarthritis who have not improved with standard treatments receive one of these injections into the knee joint as part of their usual care. Eye pressure in both eyes is measured before the injection and one week later. By comparing the change in eye pressure between the two steroid groups, the study aims to better understand the risk of steroid-related increases in eye pressure and to help doctors choose safer treatment options, especially for patients who may be at risk for glaucom

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic early-stage knee osteoarthritis Patients aged 18-75 years No prior eye surgery No history of elevated IOP or glaucoma diagnosis Patients not receiving any medical treatment altering IOP

Exclusion Criteria:

* IOP >21 mm Hg Patients with a previous or current diagnosis of glaucoma Patients aged <18 and >75 years History of or ongoing ocular disease Use of medications (oral CSs, diazoxide, etc.) altering IOP

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-10-02 (Actual); Primary Completion 2025-11-02 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Change in Intraocular Pressure (IOP) From Baseline to 1 Week | Baseline (before intra-articular steroid injection) and 1 week after injection
  ntraocular pressure (IOP) in both eyes will be measured in mmHg using noncontact tonometry at baseline (before the intra-articular injection) and 1 week after the injection. Change in IOP (ΔIOP) will be calculated for each eye as the value at 1 week minus the baseline value. The primary outcome is the mean change in IOP in each treatment group

CONTACTS AND LOCATIONS:
Locations (1):
- Niğde Ömer Halisdemir University, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided